CLINICAL TRIAL: NCT01036048
Title: Drug Eluting Stents Versus Bare Metal Stents in Saphenous Vein Graft Disease: Insights From a Meta-analysis
Brief Title: A Meta-analysis of Drug Eluting Stents Versus Bare Metal Stents in Saphenous Vein Graft Disease
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: navarese, Catholic University of the Sacred Heart
Other Study IDs: N28LBCF80-07
Record Dates: First submitted 2009-12-07; First posted 2009-12-21 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Saphenous Vein Graft Disease
Keywords: saphenous vein graft; stent
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cabg disease: pts with saphenous vein graft disease
  Interventions: Device: drug eluting stent; Device: bare metal stent

INTERVENTIONS:
Device: drug eluting stent — pts with cabg disease treated with drug eluting stent
  Other Names: des
Device: bare metal stent — pts with cabg disease treated with bare metal stent
  Other Names: bms

SUMMARY:
A meta-analysis to compare outcomes of drug eluting stents (DES) versus bare metal stent (BMS) in saphenous vein graft (SVG) disease.

DETAILED DESCRIPTION:
To compare outcomes (death, myocardial infarction, target vessel revascularization) of drug eluting stent versus bare metal stent in saphenous vein graft disease.

ELIGIBILITY:
Inclusion Criteria:

* CABG disease
* randomized studies
* not randomized studies

Exclusion Criteria:

* studies reporting composite and not single endpoints, duplicate reporting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with CABG disease
Sampling Method: Non-Probability Sample
Enrollment: 5806 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
death | years depending from studies retrieved

SECONDARY OUTCOMES:
myocardial infarction | years depending from study retrieved
target vessel revascularization | years depending from study retrieved

CONTACTS AND LOCATIONS:
Overall Officials: ALESSANDRO LUPI, MD, Principal Investigator — OSPEDALE MAGGIORE NOVARA; ELIANO NAVARESE, MD, Principal Investigator — CATHOLIC UNIVERSITY OF SACRED HEART

REFERENCES:
- [Derived] Lupi A, Navarese EP, Lazzero M, Sansa M, De Servi S, Serra A, Bongo AS, Buffon A. Drug-eluting stents vs. bare metal stents in saphenous vein graft disease. Insights from a meta-analysis of 7,090 patients. Circ J. 2011;75(2):280-9. doi: 10.1253/circj.cj-10-0186. Epub 2010 Dec 14. PMID 21173499